CLINICAL TRIAL: NCT06556238
Title: Metabolism-Informed Care to Aid Alaska Native People to Quit Smoking (QUIT): Pilot Intervention and Assessment of Barriers and Facilitators of Implementation
Brief Title: Metabolism-Informed Care to Aid Alaska Native People to Quit Smoking (QUIT)
Acronym: QUIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southcentral Foundation (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Georgia Michlig, Senior Researcher, Southcentral Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1958237; S06GM142122 (NIH)
Record Dates: First submitted 2024-08-08; First posted 2024-08-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotine Metabolite Ratio (Experimental): Subjects identified as cigarette smokers wishing to quit will receive the Nicotine Metabolite Ratio (NMR) test in a primary care setting and the results of the NMR will be used to inform medication recommendations for tobacco cessation.
  Interventions: Other: Nicotine Metabolite Ratio

INTERVENTIONS:
Other: Nicotine Metabolite Ratio — Blood specimens will be drawn, in clinic, by clinical staff trained in blood collection (e.g., certified medical assistant, nurse). Through regular clinic procedures, lab staff will ship for processing to Quest. Quest uses liquid chromatography tandem mass spectrometry with a limit of detection of 2ng/ml for all analytes and will quantify NMR within 3-6 days of sample arrival. Samples will be consumed during testing. Results of NMR will be returned to primary care providers, and NMR-informed medication recommendations will be made to participants.

SUMMARY:
The purpose of this study is to refine and pilot an intervention using the Nicotine Metabolite Ratio (NMR) to inform the selection of pharmacologic treatment to increase smoking abstinence among Alaska Native and American Indian people. This is a single-arm pilot trial to assess and improve acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

(Patients)

* Alaska Native or American Indian person by self-report
* eligible for or already receiving services at Southcentral Foundation (SCF)
* age 18 years or older
* daily smoking in the past 30-days
* if other nicotine or tobacco products are used, cigarettes are main product used
* planning to schedule an appointment with the Quit Tobacco Program to seek smoking cessation treatment in the next 30 days
* willing to make a quit attempt within 30 days of enrollment in the Quit Tobacco Program
* willing to have a blood test to inform their treatment
* willing to try a pharmacologic treatment
* willing to provide a saliva sample
* has phone service
* has access to broadband internet on mobile phone at home, work, or other location
* has an Android or iPhone mobile phone compatible with the Smokerlyzer app

(Staff)

- Staff participants of qualitative interviews to assess acceptability and feasibility of the intervention must be a health care professional at Southcentral Foundation (SCF), involved in the care of one of the participants of the study, that is their care team staff; including but not limited to: primary care providers, tobacco treatment specialists/health educators, pharmacists, nurse case managers, behavioral health consultants, certified medical assistants, and lab technicians.

Exclusion Criteria:

(Patients)

* Participated in the prior study phase
* participated in a cessation program during the past 3 months
* their provider has not approved varenicline in their referral to the Quit Tobacco Program
* has history of serious hypersensitivity or skin reactions to varenicline
* has bleeding disorder or is currently receiving cancer treatment
* questionable capacity or impaired decision-making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention implementation: Enrollment | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  Proportion of eligible persons who enroll
Feasibility of intervention implementation: Treatment recommendations | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  Proportion who use treatment recommended by NMR results
Feasibility of intervention implementation: Semi-structured interviews | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  Qualitatively, based on semi-structured interviews with a selection of participants and care team/administrators, thematic analysis will explore barriers and facilitators to using metabolism-informed care, as well as fidelity challenges in adhering to the recommended treatment.
Acceptability of metabolism-informed intervention: Quantitative | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  Mean of fourteen, 3-point, Likert-scale survey responses (agree/neither agree nor disagree/disagree, with a "prefer not to answer" option). These items will assess intervention and process acceptability including timeliness of the procedures and recommendation, composition of the team, clarity of communication, ease of understanding pilot measures, willingness to recommend, and satisfaction. These items will be combined into a summary score indicating overall acceptability of the intervention.
Acceptability of metabolism-informed intervention: Qualitative | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  Additional data will be collected qualitatively via semi-structured interviews with selected participants and care team/administrators.

SECONDARY OUTCOMES:
Smoking Cessation: Self-report | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  self-report of cigarette smoking for the past 7 days
Smoking Cessation: Expelled CO | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  expelled CO<4ppm according to a handheld breath monitor which connects to a mobile device (iCO Smokerlyzer®, Bedfont Scientific)
Smoking Cessation: Nicotine <10ng/mL | Beta phase (n=10) 6 weeks; Pilot phase (n=40) 6 weeks, 12 weeks, 26 weeks
  nicotine <10ng/mL measured by a saliva test strip (Accutest® NicAlert Saliva Collection Kit)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia J Michlig, PhD, Principal Investigator — Southcentral Foundation
Locations (1):
- Anchorage Native Primary Care Center, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No